CLINICAL TRIAL: NCT01127841
Title: Study Phase II Non-randomized Prospective Open to Assess the Combination of Rituximab, Bendamustine (RB) for Patients With Follicular Lymphoma Refractory or Relapsed After Treatment With R-chemotherapy in First Line.
Brief Title: Trial of Rituximab, Bendamustine (RB) for Patients With Follicular Lymphoma Refractory or Relapsed After Treatment With R-chemotherapy in First Line
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Grupo Oncológico para el Tratamiento y el Estudio de los Linfomas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOTEL/09-01
Record Dates: First submitted 2010-03-18; First posted 2010-05-21 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-08

CONDITIONS: Follicular Non-Hodgking´s Lymphoma Refractory or Relapsed After Treatment With R-chemotherapy in First Line.
MeSH Terms: interventions — Rituximab; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rituximab and Bendamustine (Experimental)
  Interventions: Drug: Rituximab and Bendamustine

INTERVENTIONS:
Drug: Rituximab and Bendamustine — Rituximab: 375 mg/m2/day, day 1 of each cycle, iv. Bendamustine: 90 mg/m2/day, days1 and 2 fo each cycle, iv.

SUMMARY:
Evaluate the effectiveness of rituximab, bendamustine (r) in terms of complete response and response complete not confirmed.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Patients with follicular lymphoma grade 1, 2 or 3a, CD20 +, histologically confirmed lymph node biopsy or tissue.
3. Follicular lymphoma patients previously treated with the combination of rituximab and chemotherapy (R-CHOP, R-CVP, R-fludarabine), having received rituximab maintenance, refractory to a first line (excluding radiotherapy) or relapsed after having achieved any response to previous treatment.
4. ECOG ≤ 2.
5. Signed written informed consent

Exclusion Criteria:

1. Clinical suspicion or documentation of histological transformation.
2. Patients with hypersensitivity to rituximab.
3. Prior autologous or allogeneic transplant.
4. CNS infiltration by LF (primary CNS lymphoma or lymphomatous meningitis).
5. Past or active Hepatitis B (at least one of the following markers HBsAg, HBe Ag, anti-HBc, HBV DNA).
6. HCV infection. HIV infection or other conditions of severe immunosuppression.
7. Previous neoplasms except non-melanoma skin cancer of the cervix or adequately treated.
8. Congestive heart failure> NYHA grade 1.
9. Impaired renal function (creatinine> 1.5 x Upper Limit of Normal, ULN) or creatinine clearance <50 ml / h, not related to lymphoma.
10. Impaired liver function (bilirubin, AST / ALT or GGT> 2 x ULN) were not related to lymphoma.
11. Women who are nursing or pregnant.
12. Patients with heart disease, pulmonary, neurological, psychiatric or severe metabolic and not secondary to lymphoma.
13. Severe acute or chronic infection in activity.
14. Any other concurrent medical or psychological comorbidity that might interfere with participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-07; Primary Completion 2013-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
the primary endpoint is the complete response and unconfirmed complete response according to the criteria of the International Workshop to Standardize Response Criteria for NHL | Four years
  Evaluation of response to induction treatment at 6 months after inclusion of the patient. Evaluation of response to maintenance treatment at 2 years after finishing the induction treatment.

SECONDARY OUTCOMES:
Secondary endpoint included an assessment of the following parameters:Global Survival,progression-Free survival,Disease-Free Survival,Duration of the Response. | Four years

CONTACTS AND LOCATIONS:
Locations (18):
- Spain (18):
  - Hospital G. U. de Alicante, Alicante, Alicante
  - Hospital de Elche, Elche, Alicante
  - Hospital Insular de Gran Canarias, Canarias, Canary Islands
  - Hospital U. de Gran Canarias Dr. Negrín, Canarias, Canary Islands
  - Hospital uan Ramón Jiménez, Huelva, Huelva
  - Hospital San Pedro de La Rioja, Logroño, La Rioja
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Costa del Sol, Marbella, Malaga
  - Hospital Son Dureta, Mallorca, Mallorca
  - Complejo Hospitalario de Pontevedra, Pontevedra, Pontevedra
  - Instituto Oncologico de San Sebastian, Donostia / San Sebastian, San Sebastian
  - Hospital Virgen de la Macarena, Seville, Sevilla
  - Hospital Sant Joan de Reus, Reus, Tarragona
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Tenerife
  - Hospital Virgen de la Salud, Toledo, Toledo
  - Hospital General de Valencia, Valencia, Valencia
  - Hospital Universitario La Fe, Valencia, Valencia
  - Hospital Universitario Virgen de la Victoria, Málaga